Athens, 23.04.2025

Research protocol CBT

The effectiveness and efficacy of the combination of pharmacotherapy and

cognitive behavioral psychotherapy under the recovery perspective for patients

with anxiety disorders, depressive disorders, PTSD, obsessive-compulsive

disorders, personality disorders, bipolar disorders, schizophrenia and

psychotic disorders.

Dr. phil., Dipl.-Psych., Stavroula Rakitzi

Clinical psychologist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

2111180571

6989766935

Stavroula@Rakitzi.onmicrosoft.com

Description linkedin Stavroula Rakitzi

ORCID: http://0000-0002-5231-6619

Polyxeni Georgila, M. D. Psychiatrist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

6932905259

polyxenigeorgila@gmail.com

Description linkedin Polyxeni Georgila

ORCID: http://0000-0003-3137-506X

1

Cognitive behavioral psychotherapy presents evidence-based psychotherapy and is

one of the most effective psychotherapies today for all mental health disorders. Many

studies are published.

The combination of pharmacotherapy and cognitive behavioral psychotherapy is one

of the most frequent treatments that we offer in our private practice. The recovery

perspective, the combination of objective and subjective recovery plays an important

role in our treatment. We would like to research the effectiveness and efficacy of

pharmacotherapy in combination with individual CBT by anxiety disorders, depressive

disorders, obsessive compulsive disorders, bipolar disorders, schizophrenia and

psychotic disorders and personality disorders.

Study population

The outpatients from our private practice. Selection criteria:

Inclusion criteria: age 18-65, IQ ≥ 80, diagnosis anxiety disorders, depression,

obsessive-compulsive disorders, PTSD, personality disorders, bipolar disorders,

schizophrenia and psychotic disorders.

Exclusion criteria: Substance abuse and head injury.

**Compliance with ethical standards** 

Prior to the study's inclusion, the patients will read and sign written informed consent

2

for their involvement in this research project. Information that could reveal the patients' identities was left out. The authors adhere to the APA ethical standards.

Scientists who treat patients in private practices are not prohibited by Greek authorities from undertaking research projects. Private sector scientists' research efforts are not reviewed by an ethical body.

## Measures

Reliable and valid tests are going to be administered before the therapy, after the therapy and in a follow-up after 6 months after therapy.

Aster et al. (2006) should be used before treatment to show the burden of cognitive dysfunction and intellectual ability, and it is repeatable after one year. An intelligence quotient (IQ) ≥ 80 is a necessary condition to participate in therapy. The Positive and Negative Syndrome Scale (PANSS) (Kay et al., 1987; Lykouras et al., 2005), WHODAS 2 0 (Koumpouros et al., 2018; WHO, 2001) for disability and functional capacity, the Recovery Assessment Scale-Domains and Stages (RAS-DS) (Hancock et al., 2019, 2023) for the evaluation of the recovery process and clinical global impression scale (CGI) for the evaluation of the global functioning (Busner & Targum, 2007; Guy, 1976) The symptom checklist 90-R (Donias et al., 1991), the Altman self-rating Mania Scale

(Altman et al., 1997) (Greek Version), the Young Mania Rating Scale (Young et al., 1978), the Symptoms Rating Scale for Depression and Anxiety (SRSDSA) (Bech, 1993; Fountoulakis, 2003), the Hamilton Depression Scale (HAM-D) (Hamilton, 1960) (the Greek version), the Montgomery and Asperg Depression Rating Scale (MADRS) (Montgomery & Asperg, 1979; Williams & Kobak, 2008) (the Greek version) and the psychotic symptom rating scales (PSYRATS) (Haddock, 1999) can also be used.

The project will begin in May 2025 and finish in December 2027.

## Statistical analysis

A GLM and regression analysis should be performed to see if the therapy groups which receive pharmacotherapy and CBT are improved after the therapy and in a follow-up after 6 months. Effect sizes will also be computed.

## References

- 1. Altman, E.G., Hedecker, D., Peterson, J.L., & Davis M. (1997). The Altman self rating mania scale. Biological Psychiatry, 42, 948-955.
  - 2. Aster, M., Neubauer, M., & Horn R. (2006) Wechsler-Intelligenztest für Erwachsene WIE. Frankfurt: Harcourt Test Services.
  - 3. Bech, P. (1993). Rating scales for Psychopathology, Health Status and Quality
  - of Life. Berlin, Heidelberg, New York: Springer-Verlag.
  - 4. Busner, J., & Targum, S.D. (2007). The Clinical Global Impressions Scale. Applying a research tool in clinical practice. Psychiatry, 29-37.
- 5. Donias, S., Karastergiou, A., & Manos N. (1991). Standardization of the symptom checklist-90-R rating scale in a Greek population. Psychiatriki, 2(1), 42-48.
  - 6. Fountoulakis, K.N., Iacovides, A., Kleanthous, S., Samolis, S., Gougoulias, K.,
  - Kaprinis GSt., & Bech, P. (2003). The Greek translation of the symptoms rating scale for depression and anxiety: preliminary results of the validation study. BMC Psychiatry, 3, 21. http://www.biomedcentral.com/1471-244X/3/21.
  - 7. Guy, W. (ed). (1976). ECDEU Assessment. Manual for Psychopharmacology.
  - Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration, 1976.
  - 8. Haddock, G., McCarron, J., Tarrier, N., Faragher, E.B. (1999). Scales to measure dimensions of hallucinations and delusions: the psychotic symptom

rating scales (PSYRATS). Psychological Medicine, 29(4), 879-889.

9. Hancock, N., Scanlan, J.N., Bundy, A.C., Honey, A. (2019). Recovery Assessment Scale –Domains & Stages (RAS-DS) Manual- Version 3. Sydney: University of Sydney.

10.Hancock, N., & the University of Sydney (2023). Rakitzi S. Katoudi S. Recovery

Assessment Scale-Domains & Stages (RAS-DS). The Greek version.

11.Kay, S.R., Fiszbein, A., & Opler LA. (1987). The positive and negative syndrome scale (PANSS) for schizophrenia. Schizoprenia Bulletin, 13(2), 261-276.

12.Kosmidou, M., & Vlahou, Ch. (2010). The Greek verbal memory test. Athens:

Parisianos.

13.Koumpouros, Y., Papageorgiou, E., & Sakellari E. et al. (2018). Adaptation and

psychometric properties evaluation of the Greek version of WHODAS 2.0. Pilot application in Greek elderly population. Health Services and Outcomes Research Methodology, 18(1), 63-74. https://doi.org/10.1007/s10742-017-0176-x

14.Lykouras, L., Botsis, A., & Oulis P. (2005). The PANSS Scale. Athens: Scientific

Publications.

15.Montgomery, S. A., & Asberg, M. (1979). A new depression scale designed to

be sensitive to change. British Journal of Psychiatry, 134(4),382-389.

- 16. Rakitzi, S. (2023). Clinical psychology and cognitive behavioral psychotherapy. Recovery in mental health. Springer.
- 17. Williams, J.B.W., & Kobak, K. A. (2008). Development and reliability of a structured interview guide for the Montgomery-Asberg Depression Rating Scale (SIGMA). The British Journal of Psychiatry, 192(1), 52-58.

18. World Health Organization. International classification of functioning, disability

and health (ICF). Geneva: World Health Organization; 2001.

19. Young, R.C., Biggs, J.T., Ziegler V.E., & Meyer, D.A. (1978). A rating scale for

mania: reliability, validity and sensitivity. British Journal of Psychiatry, 133, 429-435.